CLINICAL TRIAL: NCT04637139
Title: An Open Label Phase 1 Study in Healthy Adult Male Subjects to Determine the Mass Balance Recovery, Absorption, Metabolism, and Excretion of [14C] Vebicorvir Following Single Oral Dose Administration
Brief Title: A Study to Evaluate the Mass Balance Absorption and AME of VBR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI H0731 108
Record Dates: First submitted 2020-10-30; First posted 2020-11-19 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Chronic Hepatitis B
Keywords: CHB; HBV; hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): VBR 300 mg solution containing 2 µCi [14C]VBR
  Interventions: Drug: Vebicorvir (VBR)

INTERVENTIONS:
Drug: Vebicorvir (VBR) — 300mg Vebicovir containing 2 µCi [14C]VBR.

SUMMARY:
This Phase 1 Study will determine the mass balance recovery, absorption, metabolism, and excretion of [14C] Vebicorvir in healthy male subjects

ELIGIBILITY:
* Consent
* Male between 18 and 55 years of age (inclusive) at the time of Screening
* Body mass index (BMI) between ≥18.0 kg/m2 and ≤32.0 kg/m2 at Screening; body weight between ≥55.0 kg and ≤100.0 kg at Screening
* Considered to be in good health by the Investigator

Exclusion Criteria:

* History or presence of any condition (e.g., chronic diarrhea) or prior surgery (e.g., gastric bypass)
* Clinically significant abnormal medical history
* History of cancer that has not been in full remission for >5 years
* Acute illness within 14 days prior to study drug administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Mass Balance: Cumulative Amount of [14C] Radiolabel Excreted in Urine up to the Last Sampling Interval (Ae-urine, 14C) | Before dosing and at prespecified time intervals up to 168 hours after dosing
Mass Balance: Cumulative Amount of [14C] Radiolabel Excreted in Feces up to the Last Sampling Interval (Ae-feces, 14C) | Before dosing and at prespecified time intervals up to 168 hours after dosing

SECONDARY OUTCOMES:
Number of Participants with One or More Adverse Events | Up to 168 hours
Number of Participants Discontinued from the Study Due to an Adverse Event | Up to 168 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided